CLINICAL TRIAL: NCT04960462
Title: Case Report of Nerve Root Sleeve Reinforcement and Reconstruction and Sacral Canal Plasty for the Treatment of Sacral Canal
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018064
Record Dates: First submitted 2021-07-04; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2017-01

CONDITIONS: Tarlov Cysts
Keywords: tarlov cysts surgery
MeSH Terms: conditions — Tarlov Cysts

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the treatment of sacral cysts in patients with sacral cysts by using nerve root sleeve reinforcement: The clinical data of patients with sacral cysts treated with nerve root sleeve reinforcement and reconstruction of the sacral canal cyst were summarized and followed up from 3 to 6 months after the operation to form a case summary and report.
  Interventions: Procedure: nerve root sleeve reinforcement

INTERVENTIONS:
Procedure: nerve root sleeve reinforcement — treatment of sacral cysts in patients with sacral cysts by using nerve root sleeve reinforcement

SUMMARY:
A retrospective study of the changes in the VAS scores and imaging examinations after the reconstruction and reinforcement of nerve root sleeves and caudal angioplasty for the treatment of sacral cysts from August 2017 to January 2018 was used to evaluate the efficacy of the surgical prescription.

DETAILED DESCRIPTION:
Objective: To clarify the curative effect of nerve root sleeve reconstruction and reinforcement and caudal plasty in the treatment of sacral cysts Design: A retrospective study of the changes in the VAS score and imaging examinations after the reconstruction and reinforcement of nerve root sleeves and sacral canoplasty for the treatment of sacral cysts from August 2017 to January 2018 to evaluate the efficacy of the surgical prescription.

ELIGIBILITY:
Inclusion Criteria:a) Symptomatic nerve root cyst diagnosed by MRI b) The capsule of the cyst is intact and the sacral lamina is not defective c) No other diseases of the nervous system, pelvic floor and important organs d) Reconstruction of patients with artificial dural nerve root sleeve reinforcement -

Exclusion Criteria:a) Non-radiotomy cyst or asymptomatic cyst b) The cyst causes severe bone erosion to lamina absorption c) Combined with other diseases of the nervous system, pelvic floor and important organs d) Those who have not used artificial dura mater for nerve root sleeve reinforcement and reconstruction

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical data (symptoms, signs, imaging findings) of patients with sacral cysts treated with sacral cyst reconstruction using nerve root sleeve reinforcement
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Symptomatic nerve root cyst diagnosed by MRI | 2017/08-2018/01
  The capsule of the cyst is intact and the sacral lamina is not defective
  ,No other diseases of the nervous system, pelvic floor and important organs Reconstruction of patients with artificial dural nerve root sleeve reinforcement

CONTACTS AND LOCATIONS:
Overall Officials: bin liu, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No